CLINICAL TRIAL: NCT00266968
Title: Assessment of the Outcomes of Children With Congenital Single Ventricle Heart
Brief Title: Outcomes of Children With Congenital Single Ventricle Heart
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Chairman, Children's Healthcare of Atlanta Institutional Review Board
Other Study IDs: 03-005
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; single ventricle
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Univentricular Heart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Congenital heart disease affects 1 in 100 newborn babies each year and more than 2,000,000 Americans have a congenital heart defect. One common defect treated at Children's Healthcare of Atlanta at Egleston is single ventricle heart. Due to these overwhelming numbers, the use of diagnostic imaging technology to assess these defects and heart function is an important step in the evolving care of this patient group.

DETAILED DESCRIPTION:
The definition of single ventricle can mean a ventricle that is hypoplastic, too small, or completely absent. Either the right or left ventricle may be affected. There may also be other cardiac anomalies present. Infants with a single ventricle develop distress after birth when the ductus arteriosus and foramen ovale close. This may happen within hours or days of delivery. The severity of symptoms is determined by the degree of defect. But, single ventricle patients will not survive without treatment. Patients with only one functioning ventricle can usually expect either a heart transplant or a series of palliative surgeries or sometimes both. Their care is very complex requiring a team of dedicated practitioners to manage drug therapy, medical support and surgery.

At Children's Healthcare of Atlanta at Egleston, it is standard of care for a patient with a single ventricle heart to undergo many non-invasive imaging studies and sometimes invasive studies such as heart catheterization. Results of the studies provide valuable information used for treatment decisions and evaluation of heart function. We propose to do a retrospective chart review of patient data including a review of their invasive and non-invasive studies.

ELIGIBILITY:
Inclusion Criteria:

* Single Ventrical heart

Exclusion Criteria:

* those patients who do not have single ventrical heart

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: subjects seen at Children's Healthcare of Atlanta with single ventrical heart
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2000-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
We propose to do a retrospective chart review of patient data including a review of their invasive and non-invasive studies. | 13 years
  We propose to do a retrospective chart review of patient data including a review of their invasive and non-invasive studies.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Cuadrado, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States